CLINICAL TRIAL: NCT05653817
Title: A Multicenter Clinical Study of Carralizumab Combined With Albumin Paclitaxel and Apatinib Mesylate in the Second-line Treatment of Advanced or Metastatic Cholangiocarcinoma
Brief Title: Advanced or Metastatic Cholangiocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XJTU1AF2021LSK-062
Record Dates: First submitted 2022-12-09; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Albumin-Bound Paclitaxel; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced or metastatic cholangiocarcinoma (Experimental): A multicenter clinical study of carralizumab combined with albumin paclitaxel and apatinib mesylate in the second-line treatment of advanced or metastatic cholangiocarcinoma.Albumin-bound paclitaxel 125 mg/m2 d1,8; Carrilizumab 200mg Q3W d1; Apatinib mesylate tablet treatment: 250mg orally, once a day, continuous administration. Treatment continued or was evaluated every 2 cycles until disease progression or toxic side effects of patient intolerance to the treatment regimen.
  Interventions: Drug: Carrilizumab; Drug: Albumin-bound paclitaxel; Drug: Apatinib

INTERVENTIONS:
Drug: Carrilizumab — Carrilizumab 200mg Q3W d1
Drug: Albumin-bound paclitaxel — Albumin-bound paclitaxel 125 mg/m2 d1,8
Drug: Apatinib — Apatinib mesylate tablets for treatment: 250mg

SUMMARY:
This is a single-arm, open, multicenter trial of carralizumab in combination with albumin paclitaxel and apatinib mesylate for the second-line treatment of patients with advanced or metastatic cholangiocarcinoma. The study enlists patients with histopathologically or cytologically confirmed unresectable, recurrent, or metastatic cholangiocarcinoma (including intrahepatic, extrahepatic, and distal cholangiocarcinoma). Previously, she had received systematic internal medicine anti-tumor therapy with gemcitabine regimen as standard, which met the inclusion criteria of this study. She was given oral therapy with albumin binding paclitaxel combined with carrilizumab and apatinib mesylate. Treatment continued or was evaluated every 2 cycles until disease progression or toxic side effects of patient intolerance to the treatment regimen. To evaluate progression-free survival (PFS) in second-line therapy with carrilizumab in combination with albumin paclitaxel and apatinib mesylate in patients with advanced or metastatic cholangiocarcinoma.

DETAILED DESCRIPTION:
Cholangiocarcinoma (CCA) is a cancer that easily invades adjacent structures. Vascular endothelial growth factor (VEGF) and VEGF receptor 2 (VEGFR2) are increased in most types of cancer and inhibit tumor progression by blocking VEGF/VEGFR2 [16]. Apatinib is a highly selective VEGFR2 antagonist that inhibits apoptosis and growth of CCA cells. Apatinib is also a derivative of PTK787, and its targets include VEGFR-1, VEGFR-2, PDGFR, c-kit, c-Src, etc. The activity of Apatinib against VEGFR-2 is 137 times that of PTK787, the IC50 is only 1nmol/L, and it can strongly inhibit tumor angiogenesis. At the same time, it can also inhibit the downstream signal transduction mediated by KDR and inhibit tumor growth.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced, pathologically unresectable or metastatic bile duct epithelial cell carcinoma;
2. Previously received a chemotherapy regimen (including gemcitabine) anti-tumor systemic therapy, but did not use albumin binding paclitaxel;
3. Age ≥18 years old and under 75 years old;
4. Predicted survival ≥3 months;
5. ECOG score 0-1;
6. Child-Pugh score<8
7. There was at least one measurable tumor lesion with a long diameter ≥10 mm and a short diameter ≥15 mm on spiral CT. For general CT or physical examination, the maximum diameter must be ≥20mm;
8. The results of liver and kidney function and blood routine examination within 1 week before enrollment were consistent with the following conditions， ANC≥1.5×10^9/L,PLT≥80×10^9/L,HGB≥80g/L,Cr≤1.5×ULN,TBIL≤2.5×ULN,ALP≤2.5×ULN,AST≤2.5×ULN,ALT≤2.5×ULN
9. Patients participate voluntarily and sign informed consent forms

Exclusion Criteria:

1. Known to be severely allergic to carrilizumab, apatinib, and albumin paclitaxel;
2. Obstructive jaundice cannot be achieved 2.5×ULN after surgical intervention;
3. Patients with biliary obstruction that may occur or worsen within 4 to 6 weeks;
4. Patients with obvious coagulation mechanism disorder, active bleeding and bleeding tendency;
5. History of other malignancies within 5 years (fully treated basal cell carcinoma of the skin, out-of-situ cervix);
6. Interstitial pneumonia or pulmonary fibrosis;
7. Uncontrollable pleural effusion or ascites;
8. Severe uncontrolled medical disease, acute infection, recent history of myocardial infarction (within 3 months);
9. Pregnant or lactating mothers who refused to use appropriate contraceptive methods during the course of this study;
10. The researchers determined that the patients were not suitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-31 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 24month
  Progression-free survival

SECONDARY OUTCOMES:
OS | 24month
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: enxiao li, PHD, Principal Investigator — First hospital of Xi'an Jiaotong University